CLINICAL TRIAL: NCT03540316
Title: Treatment Outcome of Short Implant Assisted Mandibular Overdenture in Combination With Low Level Laser Therapy
Brief Title: Treatment Outcome of Short Implant Assisted Mandibular Overdenture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sara Zayed (Other)
Responsible Party: Sponsor-Investigator, Sara Zayed, Director, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 01032018
Record Dates: First submitted 2018-05-02; First posted 2018-05-30 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Atrophy of Edentulous Mandibular Alveolar Ridge
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Two short implants and 2 minutes LLLT (Active Comparator): Patients receiving 2 short dental implants assisted mandibular over-denture and Low level laser therapy (LLLT) for 2 minutes .
  Interventions: Combination Product: Two short implants and 2 minutes LLLT
- Two short implants and 4 minutes LLLT (Active Comparator): Patients receiving 2 short dental implants assisted mandibular over-denture and LLLT for 2 minutes .
  Interventions: Combination Product: Two short implants and 4 minutes LLLT
- Four short implants and 2 minutes LLLT (Active Comparator): Patients receiving 4 short dental implants assisted mandibular over-denture and LLLT for 2 minutes .
  Interventions: Combination Product: Four short implants and 2 minutes LLLT
- Four short implants and 4 minutes LLLT (Active Comparator): Patients receiving 4 short dental implants assisted mandibular over-denture and LLLT for 4 minutes .
  Interventions: Combination Product: Four short implants and 4 minutes LLLT

INTERVENTIONS:
Combination Product: Two short implants and 2 minutes LLLT — Patients with edentulous atrophied mandibular ridge will receive 2 short dental implants and LLLT for 2 minutes.
  Arms: Two short implants and 2 minutes LLLT
Combination Product: Two short implants and 4 minutes LLLT — Patients with edentulous atrophied mandibular ridge will receive 2 short dental implants and LLLT for 4 minutes.
  Arms: Two short implants and 4 minutes LLLT
Combination Product: Four short implants and 2 minutes LLLT — Patients with edentulous atrophied mandibular ridge will receive 4 short dental implants and LLLT for 2 minutes.
  Arms: Four short implants and 2 minutes LLLT
Combination Product: Four short implants and 4 minutes LLLT — Patients with edentulous atrophied mandibular ridge will receive 4 short dental implants and LLLT for 4 minutes.
  Arms: Four short implants and 4 minutes LLLT

SUMMARY:
This study evaluates the use of short dental implants to support mandibular overdenture together with the use of laser therapy for treatment of patients with atrophic ridges. All participants will receive laser therapy; half of participants will receive two short implants and the other half will receive four short implants.

DETAILED DESCRIPTION:
The conventional solution to complete edentulism is the use of complete removable dentures. One negative effect of edentulism is resorption of the edentulous ridge over time. Construction of a successful mandibular complete denture for patients with advanced mandibular ridge resorption is often difficult and on some occasions virtually impossible. It has been proved that when implants are placed, bone gets stimulated resulting in minimal bone loss. But anatomic limitations to implant placement have been observed in atrophic ridges, so short implants introduced as a recent alternative to aggressive surgical procedures proposed to compensate for tissue deficiency. Also, Low Level Laser Therapy (LLLT) has proven success in improving implant stability which is very crucial in short implants. Thus, the purpose of this study is to evaluate and compare the treatment outcome of mandibular overdenture assisted by two short implants versus that assisted by four short implants in combination with LLLT.

ELIGIBILITY:
Inclusion Criteria:

* Completely edentulous patients.
* Patients with mandibular resorbed edentulous ridge.
* Medically fit patients with no systemic conditions.
* Class I ridge relation.
* Adequate zone of keratinized mucosa.

Exclusion Criteria:

* Metabolic bone disease or unstable systemic condition.
* Heavy smokers.
* A history of radiotherapy in the head and neck region.
* Physical or mental disability.
* Temporomandibular and neuromuscular disorders.

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of changes in implant stability (Implant Stability Quotient). | Baseline, 6 months &12 months.
  Implant stability can be defined as the absence of clinical mobility. It will be assessed at the time of implant placement (baseline) ,then six months and twelve months later, by the resonance frequency analysis using Osstel devise which measure implant oscillation frequency on the bone;Implant Stability Quotient (ISQ) .

SECONDARY OUTCOMES:
Peri-implant marginal bone changes. | Baseline, 6 months &12 months.
  Radiographic assessment of bone level changes around each implant will be performed to detect peri-implant crestal bone changes using standardised digital periapical x-ray. It will be assessed at the time of implant placement, six months and twelve months later.
Assessment of changes in peri-implant probing depth . | Baseline, 6 months &12 months.
  Peri-implant probing depth is the distance between the gingival margin and the most apically probeable portion, in millimetres. It will be measured at four sites of each implant (mesially, labially, distally, lingually) by using a graduated periodontal probe which will be held parallel to the long axis of the implant and introduced to the peri-implant sulcus till there is slight resistance. The mean record for each implant will be calculated. It will be evaluated at time of definitive prosthesis insertion then, six months and twelve months after implant placement.
Assessment of changes in modified gingival index | Baseline, 6 months &12 months.
  To qualify the degree of peri-implant inflammation, the modified gingival index will be used. It will be measured at four sites around each implant (mesially, labially, distally, lingually) and the mean record for each implant will be calculated. It will be evaluated at time of definitive prosthesis insertion, then six months and twelve months after implant placement.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Zayed, Study Director — Alexandria University
Locations (1):
- Faculty of dentistry, Alexandria, Egypt

REFERENCES:
- [Background] Thomason JM, Feine J, Exley C, Moynihan P, Muller F, Naert I, Ellis JS, Barclay C, Butterworth C, Scott B, Lynch C, Stewardson D, Smith P, Welfare R, Hyde P, McAndrew R, Fenlon M, Barclay S, Barker D. Mandibular two implant-supported overdentures as the first choice standard of care for edentulous patients--the York Consensus Statement. Br Dent J. 2009 Aug 22;207(4):185-6. doi: 10.1038/sj.bdj.2009.728. PMID 19696851
- [Background] Maniewicz S, Buser R, Duvernay E, Vazquez L, Loup A, Perneger TV, Schimmel M, Muller F. Short Dental Implants Retaining Two-Implant Mandibular Overdentures in Very Old, Dependent Patients: Radiologic and Clinical Observation Up to 5 Years. Int J Oral Maxillofac Implants. 2017 Mar/Apr;32(2):415-422. doi: 10.11607/jomi.5361. PMID 28291859
- [Background] Mandic B, Lazic Z, Markovic A, Mandic B, Mandic M, Djinic A, Milicic B. Influence of postoperative low-level laser therapy on the osseointegration of self-tapping implants in the posterior maxilla: a 6-week split-mouth clinical study. Vojnosanit Pregl. 2015 Mar;72(3):233-40. doi: 10.2298/vsp131202075m. PMID 25958474
- [Background] Malo P, de Araujo Nobre M, Rangert B. Short implants placed one-stage in maxillae and mandibles: a retrospective clinical study with 1 to 9 years of follow-up. Clin Implant Dent Relat Res. 2007 Mar;9(1):15-21. doi: 10.1111/j.1708-8208.2006.00027.x. PMID 17362493
- [Derived] Zayed SM, Noureldin MG. Rehabilitation of Atrophic Mandible with Ultrashort Implants Combined with Photobiomodulation Therapy: A Split-Mouth Design Study. Saudi J Med Med Sci. 2022 Sep-Dec;10(3):198-206. doi: 10.4103/sjmms.sjmms_635_21. Epub 2022 Aug 22. PMID 36247059